CLINICAL TRIAL: NCT01257204
Title: A Phase 2B Pilot Study of Short-Term Treatment of BMS-790052 in Combination With Peg-Interferon Alfa-2a and Ribavirin in Treatment Naive Subjects With Chronic Hepatitis C Genotype 2 or 3 Infection
Brief Title: Study in Genotype 2 or 3 Patients With Chronic Hepatitis Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AI444-031; 2010-022408-28 (EudraCT Number)
Record Dates: First submitted 2010-12-01; First posted 2010-12-09 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-11

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): Placebo + Pegylated interferon alfa-2a + Ribavirin
  Interventions: Drug: Placebo; Drug: Pegylated interferon alfa-2a; Drug: Ribavirin
- 12 Week Cohort (Experimental): Daclatasvir + Pegylated interferon alfa-2a + Ribavirin
  Interventions: Drug: Daclatasvir; Drug: Pegylated interferon alfa-2a; Drug: Ribavirin
- 16 Week Cohort (Experimental): Daclatasvir + Pegylated interferon alfa-2a + Ribavirin
  Interventions: Drug: Daclatasvir; Drug: Pegylated interferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Placebo — Tablets, oral, 0 mg, once daily, for 24 weeks
  Arms: Control
Drug: Daclatasvir — Tablets, oral, 60 mg, once daily, for 12, 16, or 24 weeks
  Other Names: BMS-790052
  Arms: 12 Week Cohort; 16 Week Cohort
Drug: Pegylated interferon alfa-2a — Solution for injection, subcutaneous injection, 180 µg/0.5 mL, once weekly, for 12, 16, or 24 weeks
  Other Names: Pegasys®
Drug: Ribavirin — Tablets, oral, 800 mg, twice daily, for 12, 16, or 24 weeks
  Other Names: Copegus®

SUMMARY:
To identify a shorter duration of antiviral therapy (12 or 16 weeks) for the combination of daclatasvir with pegylated interferon alfa-2a and ribavirin.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants chronically infected with hepatitis C virus (HCV) genotype 2 or 3
* No previous exposure to an interferon formulation (ie, interferon alfa, pegylated interferon alfa-2a ) or ribavirin
* Body mass index (BMI) of 18 to 35 kg/m^2, inclusive. BMI=weight (kg)/height (m)^2
* Males and females, 18 - 70 years of age

Key Exclusion Criteria:

* Liver transplant recipients
* Documented or suspected hepatocellular carcinoma
* Evidence of decompensated cirrhosis
* History of chronic hepatitis B virus (HBV). Patients with resolved HBV infection may participate
* Current or known history of cancer
* Any gastrointestinal disease or surgical procedure that may impact the absorption of study drug
* Inability to tolerate oral medication
* Poor venous access
* Severe psychiatric disease
* History of chronic pulmonary disease
* History of cardiomyopathy, coronary artery disease (including angina), interventive procedure for coronary artery disease (including angioplasty, stent procedure, or cardiac bypass surgery), ventricular arrhythmia,, or other clinically significant cardiac disease
* History of or current electrocardiogram findings indicative of cardiovascular instability
* Preexisting ophthalmologic disorders considered clinically significant on eye
* History of uncontrolled diabetes mellitus
* Any known contraindication to pegylated interferon alfa-2a or ribavirin not otherwise specified.
* Positive hepatitis B virus surface antigen, HIV-1 or HIV-2 Ab
* Prior exposure to any HCV direct antiviral agent (eg, HCV protease, polymerase, previous nonstructural protein 5A inhibitors)
* Exposure to any investigational drug or placebo

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2010-12; Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (26):
- United States (4):
  - California Liver Institute, Los Angeles, California
  - Digestive Disease Associates, P.A., Baltimore, Maryland
  - Options Health Research, Llc, Tulsa, Oklahoma
  - Alamo Medical Research, San Antonio, Texas
- Australia (6):
  - Local Institution, Darlinghurst, New South Wales
  - Local Institution, Westmead Nsw, New South Wales
  - Local Institution, Adelaide, South Australia
  - Local Institution, Clayton Vic, Victoria
  - Local Institution, Fremantle, Western Australia
  - Local Institution, Camperdown
- Canada (6):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Toronto, Ontario
- Local Institution, Hvidovre, Denmark
- France (6):
  - Local Institution, Créteil
  - Local Institution, Lille
  - Local Institution, Montpellier
  - Local Institution, Nice
  - Local Institution, Paris
  - Local Institution, Pessac
- Italy (3):
  - Local Institution, Brescia
  - Local Institution, Cisanello (pisa)
  - Local Institution, Viale Del Policlinico, 155

REFERENCES:
- [Derived] Dore GJ, Lawitz E, Hezode C, Shafran SD, Ramji A, Tatum HA, Taliani G, Tran A, Brunetto MR, Zaltron S, Strasser SI, Weis N, Ghesquiere W, Lee SS, Larrey D, Pol S, Harley H, George J, Fung SK, de Ledinghen V, Hagens P, McPhee F, Hernandez D, Cohen D, Cooney E, Noviello S, Hughes EA. Daclatasvir plus peginterferon and ribavirin is noninferior to peginterferon and ribavirin alone, and reduces the duration of treatment for HCV genotype 2 or 3 infection. Gastroenterology. 2015 Feb;148(2):355-366.e1. doi: 10.1053/j.gastro.2014.10.007. Epub 2014 Oct 13. PMID 25311593
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 196 participants were enrolled, of which 152 participants were randomized; remaining 44 participants did not meet study criteria. Of randomized participants:151 were treated; 1 participant withdrew consent.
Groups:
- Daclatasvir, 60 mg, 12-Week Cohort: Participants received daclatasvir tablets 60 mg orally, once daily, with pegylated-interferon alfa-2a (pegIFNα-2a) solution for injection 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 400 mg orally, twice daily, for up to 12 weeks.
- Daclatasvir, 60 mg, 16-Week Cohort: Participants received daclatasvir tablets 60 mg orally, once daily, with pegIFNα-2a solution for injection 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 400 mg orally, twice daily, for up to 16 weeks.
- Placebo: Participants received placebo matched with daclatasvir tablets orally, once daily, with pegIFNα-2a solution for injection 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 400 mg orally, twice daily, for up to 24 weeks.
Period: Treatment Period (up to Week 24)
Arm/Group | Daclatasvir, 60 mg, 12-Week Cohort | Daclatasvir, 60 mg, 16-Week Cohort | Placebo
Started | 50 | 50 | 51
Completed | 45 | 44 | 42
Not Completed | 5 | 6 | 9
Not completed — Lack of Efficacy | 0 | 1 | 3
Not completed — Adverse Event | 3 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Poor compliance/noncompliance | 0 | 0 | 1
Not completed — Participant's request to discontinue | 1 | 2 | 2
Period: Follow-up Period (up to Week 48)
Arm/Group | Daclatasvir, 60 mg, 12-Week Cohort | Daclatasvir, 60 mg, 16-Week Cohort | Placebo
Started | 49 (Those who completed period 1 or with detectable hepatitis C virus RNA, despite length of treatment.) | 47 (Those who completed period 1 or with detectable hepatitis C virus RNA, despite length of treatment.) | 49 (Those who completed period 1 or with detectable hepatitis C virus RNA, despite length of treatment.)
Completed | 48 | 41 | 39
Not Completed | 1 | 6 | 10
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — Lost to Follow-up | 1 | 4 | 4
Not completed — Other | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Dacalatasvir, 60 mg, 12-Week Cohort: Participants received daclatasvir tablets 60 mg orally, once daily, with pegylated-interferon alfa-2a (pegIFNα-2a) solution for injection 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 400 mg orally, twice daily, up to 12 weeks.
- Daclatasvir, 60 mg, 16-Week Cohort: Participants received daclatasvir tablets 60 mg orally, once daily, with pegIFNα-2a solution for injection 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 400 mg orally, twice daily, up to 16 weeks.
- Placebo: Participants received placebo matching with daclatasvir tablets orally, once daily, with pegIFNα-2a solution for injection 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 400 mg orally, twice daily, up to 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Dacalatasvir, 60 mg, 12-Week Cohort | Daclatasvir, 60 mg, 16-Week Cohort | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 51 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (8.42) | 47.5 (9.20) | 48.8 (9.73) | 47.9 (9.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 13 | 24 | 55
  Male | 32 | 37 | 27 | 96
Hepatitis C Virus (HCV) RNA (IU/mL) [Mean (Standard Deviation); unit: Log10 IU/mL] | 6.4 (0.82) | 6.6 (0.62) | 6.6 (0.59) | 6.5 (0.69)
HCV RNA Distribution [Number; unit: participants]
  <800,000 IU/mL | 12 | 7 | 6 | 25
  ≥800,000 IU/mL | 38 | 43 | 45 | 126
Randomization Stratum [Number; unit: participants]
  HCV Genotype 2 | 24 | 23 | 24 | 71
  HCV Genotype 3 | 26 | 27 | 27 | 80
Cirrhosis Status [Number; unit: participants]
  Absent | 43 | 43 | 41 | 127
  Present | 7 | 4 | 8 | 19
  Not Reported | 0 | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response at Follow-up Week 24 (SVR24) for Hepatitis C Virus (HCV) Genotype 2
Description: SVR24 was defined as undetectable HCV RNA (HCV RNA <lower limit of quantitation [LLOQ], target not detected [TND]) at follow-up Week 24. The LLOQ was 25 IU/mL, and <LLOQ, TND was 10 IU/mL. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Follow-up Week 24
Population: All treated participants with hepatitis C virus genotype 2.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Daclatasvir, 60 mg, 12-Week Cohort: Participants received daclatasvir tablets 60 mg orally, once daily, with pegylated-interferon alfa-2a (pegIFNα-2a) solution for injection 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 400 mg orally, twice daily, up to 12 weeks.
Arm/Group | Daclatasvir, 60 mg, 12-Week Cohort | Daclatasvir, 60 mg, 16-Week Cohort | Placebo
Number analyzed (Participants) | 24 | 23 | 24
percentage of participants | 83.3 [73.6 to 93.1] | 82.6 [72.5 to 92.7] | 62.5 [49.8 to 75.2]
Statistical Analysis 1: Comparison: Daclatasvir, 60 mg, 12-Week Cohort vs Placebo; Test type: Superiority or Other; Difference = 20.8, 80% CI 2-sided [4.9 to 36.8] — The difference in the percentage of participants with antiviral response between daclatasvir and placebo was presented with a difference estimate (daclatasvir - placebo) and 80% confidence Interval
Statistical Analysis 2: Comparison: Daclatasvir, 60 mg, 16-Week Cohort vs Placebo; Test type: Superiority or Other; Difference = 20.1, 80% CI 2-sided [3.9 to 36.3] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants Achieving Rapid Virologic Response (RVR) at Week 4 for Hepatitis C Virus (HCV) Genotype 2
Description: RVR was defined as undetectable HCV RNA (HCV RNA <lower limit of quantitation [LLOQ], target not detected [TND]) at Week 4. The LLOQ was 25 IU/mL, and <LLOQ, TND was 10 IU/mL. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Week 4
Population: All treated participants with HCV genotype 2.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Daclatasvir, 60 mg, 12-Week Cohort: Participants received daclatasvir tablets 60 mg orally, once daily, along with pegylated-interferon alfa-2a (pegIFNα-2a) solution for injection 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 400 mg orally, twice daily, up to 12 weeks.
- Daclatasvir, 60 mg, 16-Week Cohort: Participants received daclatasvir tablets 60 mg orally, once daily, along with pegIFNα-2a solution for injection 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 400 mg orally, twice daily, up to 16 weeks.
- Placebo: Participants received placebo matching with daclatasvir tablets orally, once daily, along with pegIFNα-2a solution for injection 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 400 mg orally, twice daily, up to 24 weeks.
Arm/Group | Daclatasvir, 60 mg, 12-Week Cohort | Daclatasvir, 60 mg, 16-Week Cohort | Placebo
Number analyzed (Participants) | 24 | 23 | 24
percentage of participants | 87.5 [78.8 to 96.2] | 73.9 [62.2 to 85.6] | 41.7 [28.8 to 54.6]

3. Secondary Outcome: Percentage of Participants Achieving Rapid Virologic Response (RVR) at Week 4 for Hepatitis C Virus (HCV) Genotype 3
Description: as for outcome 2
Time Frame: Week 4
Population: All treated participants with HCV genotype 3.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Daclatasvir, 60 mg, 12-Week Cohort: Participants received daclatasvir tablets 60 mg orally, once daily, along with pegylated-interferon alfa-2a (pegIFNα-2a) solution for injection 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 400 mg orally, twice daily, up to 12 week s.
Arm/Group | Daclatasvir, 60 mg, 12-Week Cohort | Daclatasvir, 60 mg, 16-Week Cohort | Placebo
Number analyzed (Participants) | 26 | 27 | 27
percentage of participants | 84.6 [75.5 to 93.7] | 74.1 [63.3 to 84.9] | 37.0 [25.1 to 48.9]

4. Secondary Outcome: Percentage of Participants Achieving Complete Early Virologic Response (cEVR) at Week 12 for Hepatitis C Virus (HCV) Genotype 2
Description: cEVR was defined as undetectable HCV RNA (HCV RNA <lower limit of quantitation [LLOQ], target not detected [TND]) at Week 12. The LLOQ was 25 IU/mL, and <LLOQ, TND was 10 IU/mL. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Week 12
Population: All treated participants with HCV genotype 2.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Daclatasvir, 60 mg, 12-Week Cohort | Daclatasvir, 60 mg, 16-Week Cohort | Placebo
Number analyzed (Participants) | 24 | 23 | 24
percentage of participants | 91.7 [84.4 to 98.9] | 82.6 [72.5 to 92.7] | 75.0 [63.7 to 86.3]

5. Secondary Outcome: Percentage of Participants Achieving Complete Early Virologic Response (cEVR) at Week 12 for Hepatitis C Virus (HCV) Genotype 3
Description: as for outcome 4
Time Frame: Week 12
Population: All treated participants with HCV genotype 3.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Dacalatasvir, 60 mg, 16-Week Cohort: Participants received daclatasvir tablets 60 mg orally, once daily, with pegIFNα-2a solution for injection 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 400 mg orally, twice daily, up to 16 weeks.
Arm/Group | Daclatasvir, 60 mg, 12-Week Cohort | Dacalatasvir, 60 mg, 16-Week Cohort | Placebo
Number analyzed (Participants) | 26 | 27 | 27
percentage of participants | 80.8 [70.9 to 90.7] | 88.9 [81.1 to 96.6] | 59.3 [47.1 to 71.4]

6. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response at Follow-up Week 12 (SVR12) for Hepatitis C Virus (HCV) Genotype 2
Description: SVR12 was defined as undetectable HCV RNA (HCV RNA <lower limit of quantitation [LLOQ], target not detected [TND]) at follow-up Week 12. The LLOQ was 25 IU/mL, and <LLOQ, TND was 10 IU/mL. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Follow-up Week 12
Population: All treated participants with HCV genotype 2.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Daclatasvir, 60 mg, 12-Week Cohort | Daclatasvir, 60 mg, 16-Week Cohort | Placebo
Number analyzed (Participants) | 24 | 23 | 24
percentage of participants | 87.5 [78.8 to 96.2] | 82.6 [72.5 to 92.7] | 70.8 [58.9 to 82.7]

7. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response at Follow-up Week 12 (SVR12) for Hepatitis C Virus (HCV) Genotype 3
Description: as for outcome 6
Time Frame: Follow-up Week 12
Population: All treated participants with HCV genotype 3.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Daclatasvir, 60 mg, 12-Week Cohort | Daclatasvir, 60 mg, 16-Week Cohort | Placebo
Number analyzed (Participants) | 26 | 27 | 27
percentage of participants | 69.2 [57.6 to 80.8] | 77.8 [67.5 to 88.0] | 51.9 [39.5 to 64.2]

8. Secondary Outcome: Number of Participants With Virologic Failure for Hepatitis C Virus (HCV) Genotype 2
Description: Virologic failure was defined as:
  1. Virologic breakthrough: confirmed >1 log10 increase in HCV RNA over nadir or confirmed RNA ≥lower limit of quantitation (LLOQ) after confirmed HCV RNA <LLOQ, target not detected (TND) while on treatment
  2. <1 log10 decrease in HCV RNA from baseline at Week 4 of treatment
  3. Failure to achieve early virologic response: <2 log10 decrease in HCV RNA from baseline and HCV RNA ≥LLOQ at Week 12 of treatment
  4. HCV RNA ≥LLOQ or <LLOQ, target detected (TD) at the end of treatment (EOT) (including early discontinuation)
  5. Relapse, defined as HCV RNA ≥LLOQ or <LLOQ, TD during follow-up, after HCV RNA <LLOQ, TND at EOT.
  The LLOQ was 25 IU/mL, and <LLOQ, TND was 10 IU/mL. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Baseline up to Week 48
Population: All treated participants with HCV genotype 2. Here, "n" signifies the number of participants evaluable for the respective category.
Measure: Number; unit: participants
Groups:
- Placebo: Participants received placebo matching with daclatasvir tablets orally, once daily, along with pegIFNα-2a solution for injection 180 mcg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 400 mg orally, twice daily, up to 24 weeks.
Arm/Group | Daclatasvir, 60 mg, 12-Week Cohort | Daclatasvir, 60 mg, 16-Week Cohort | Placebo
Number analyzed (Participants) | 24 | 23 | 24
participants
  Virologic breakthrough (n=24,23,24) | 0 | 1 | 1
  <1 log10 decrease in HCV RNA at Week4 (n=24,23,24) | 0 | 1 | 0
  HCV RNA ≥LLOQ or <LLOQ, TD at EOT (n=24,23,24) | 1 | 2 | 1
  Relapse (n=23,21,22) | 1 | 0 | 2

9. Secondary Outcome: Number of Participants With Virologic Failure for Hepatitis C Virus (HCV) Genotype 3
Description: as for outcome 8
Time Frame: Baseline up to Week 48
Population: All treated participants with HCV genotype 3. Here, "n" signifies the number of participants evaluable for the respective category.
Measure: Number; unit: participants
Arm/Group | Daclatasvir, 60 mg, 12-Week Cohort | Daclatasvir, 60 mg, 16-Week Cohort | Placebo
Number analyzed (Participants) | 26 | 27 | 27
participants
  Virologic breakthrough (n=26,27,27) | 0 | 0 | 1
  <1 log10 decrease in HCV RNA at Week4 (n=26,27,27) | 0 | 1 | 3
  HCV RNA ≥LLOQ or <LLOQ, TD at EOT (n=26,27,27) | 1 | 2 | 3
  Relapse (n=25,24,21) | 6 | 6 | 3

10. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response at Follow-up Week 24 (SVR24) for Hepatitis C Virus (HCV) Genotype 3
Description: as for outcome 1
Time Frame: Follow-up Week 24
Population: All treated participants with HCV genotype 3.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Daclatasvir, 60 mg, 12-Week Cohort | Daclatasvir, 60 mg, 16-Week Cohort | Placebo
Number analyzed (Participants) | 26 | 27 | 27
percentage of participants | 69.2 [57.6 to 80.8] | 66.7 [55.0 to 78.3] | 59.3 [47.1 to 71.4]
Statistical Analysis 1: Comparison: Daclatasvir, 60 mg, 12-Week Cohort vs Placebo; Test type: Superiority or Other; Difference = 10.0, 80% CI 2-sided [-6.8 to 26.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Daclatasvir, 60 mg, 16-Week Cohort vs Placebo; Test type: Superiority or Other; Difference = 7.4, 80% CI 2-sided [-9.4 to 24.2] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Discontinuations Due to AEs, and Treatment-related AEs and Who Died During Treatment Period
Description: AE was defined as any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not has a causal relationship with treatment. SAE was defined as a medical event that at any dose resulted in death, persistent or significant disability/incapacity, or drug dependency/abuse; was life-threatening, an important medical event, or a congenital anomaly/birth defect; or required or prolonged hospitalization. Treatment-related AE was defined as an AE that had certain, probable, possible, or unknown relationship to study drug. Mild (Grade 1): awareness of event but easily tolerated; Moderate (Grade 2): discomfort enough to cause some interference with usual activity; Severe (Grade 3): inability to carry out usual activity; Very severe (Grade 4): debilitating, significantly incapacitates participant despite symptomatic therapy. Only Grade 2-4 treatment-related AEs were reported.
Time Frame: Baseline (Day 1) up to 24 weeks (treatment period)
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Daclatasvir, 60 mg, 12-Week Cohort | Daclatasvir, 60 mg, 16-Week Cohort | Placebo
Number analyzed (Participants) | 50 | 50 | 51
participants
  AEs | 49 | 49 | 50
  SAEs | 4 | 0 | 3
  Discontinuations due to AEs | 4 | 3 | 2
  Grade 2-4 Treatment-related AEs | 27 | 22 | 30
  Deaths | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Who Died During Follow-up Period
Description: AE was defined as any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not has a causal relationship with treatment. SAE was defined as a medical event that at any dose resulted in death, persistent or significant disability/incapacity, or drug dependency/abuse; was life-threatening, an important medical event, or a congenital anomaly/birth defect; or required or prolonged hospitalization.
Time Frame: From end of treatment period up to Week 48 (follow-up period)
Population: All follow-up participants.
Measure: Number; unit: participants
Groups:
- Daclatasvir, 60 mg, 12-Week Cohort: Follow-up: Participants received daclatasvir tablets 60 mg orally, once daily, along with pegylated-interferon alfa-2a (pegIFNα-2a) solution for injection 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 400 mg orally, twice daily, up to 12 weeks during treatment period and entered into the follow-up period.
- Daclatasvir, 60 mg, 16-Week Cohort: Follow-up: Participants received daclatasvir tablets 60 mg orally, once daily, with pegIFNα-2a solution for injection 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 400 mg orally, twice daily, up to 16 weeks during treatment period and entered into the follow-up period.
- Placebo: Follow-up: Participants received placebo matching with daclatasvir tablets orally, once daily, with pegIFNα-2a solution for injection 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 400 mg orally, twice daily, up to 24 weeks during treatment period and entered into the follow-up period.
Arm/Group | Daclatasvir, 60 mg, 12-Week Cohort: Follow-up | Daclatasvir, 60 mg, 16-Week Cohort: Follow-up | Placebo: Follow-up
Number analyzed (Participants) | 49 | 47 | 49
participants
  AEs | 16 | 12 | 11
  SAEs | 2 | 0 | 0
  Deaths | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to 24 weeks (treatment period); From end of treatment period up to Week 48 (follow-up period)
Groups:
- Daclatasvir, 60 mg, 16-Week Cohort: Follow-up: Participants received daclatasvir tablets 60 mg orally, once daily, with pegIFNα-2a solution for injection 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 400 mg orally, twice daily, for up to 16 weeks during treatment period and entered into the follow-up period.
- Placebo: Follow-up: Participants received placebo matched with daclatasvir tablets orally, once daily, with pegIFNα-2a solution for injection 180 µg/0.5 mL subcutaneously, once weekly, and ribavirin tablets 400 mg orally, twice daily, for up to 24 weeks during treatment period and entered into the follow-up period.
Arm/Group | Daclatasvir, 60 mg, 12-Week Cohort | Daclatasvir, 60 mg, 16-Week Cohort | Placebo | Daclatasvir, 60 mg, 12-Week Cohort: Follow-up | Daclatasvir, 60 mg, 16-Week Cohort: Follow-up | Placebo: Follow-up
Serious Adverse Events (participants affected / at risk) | 4/50 | 0/50 | 3/51 | 2/49 | 0/47 | 0/49
Other Adverse Events (participants affected / at risk) | 49/50 | 49/50 | 48/51 | 0/49 | 0/47 | 0/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir, 60 mg, 12-Week Cohort (N=50) | Daclatasvir, 60 mg, 16-Week Cohort (N=50) | Placebo (N=51) | Daclatasvir, 60 mg, 12-Week Cohort: Follow-up (N=49) | Daclatasvir, 60 mg, 16-Week Cohort: Follow-up (N=47) | Placebo: Follow-up (N=49)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Conversion disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Adhesion (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Appendiceal Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Tonsil Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir, 60 mg, 12-Week Cohort (N=50) | Daclatasvir, 60 mg, 16-Week Cohort (N=50) | Placebo (N=51) | Daclatasvir, 60 mg, 12-Week Cohort: Follow-up (N=49) | Daclatasvir, 60 mg, 16-Week Cohort: Follow-up (N=47) | Placebo: Follow-up (N=49)
Abdominal pain (Gastrointestinal disorders) | 7 | 1 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 8 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 3 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 5 | 3 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 3 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 5 | 11 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 3 | 3 | 2 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 6 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 13 | 14 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 4 | 6 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 0 | 2 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 4 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 3 | 8 | 0 | 0 | 0
Influenza like illness (General disorders) | 10 | 9 | 7 | 0 | 0 | 0
Injection site reaction (General disorders) | 3 | 2 | 3 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 4 | 0 | 0 | 0
Asthenia (General disorders) | 6 | 7 | 7 | 0 | 0 | 0
Depression (Psychiatric disorders) | 4 | 7 | 9 | 0 | 0 | 0
Fatigue (General disorders) | 23 | 12 | 19 | 0 | 0 | 0
Injection site erythema (General disorders) | 5 | 5 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 11 | 8 | 17 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 4 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 5 | 5 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 3 | 5 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 4 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 6 | 9 | 0 | 0 | 0
Chills (General disorders) | 3 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 5 | 3 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 4 | 1 | 0 | 0 | 0
Irritability (General disorders) | 8 | 9 | 6 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 2 | 1 | 3 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 10 | 12 | 8 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 5 | 2 | 2 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 8 | 8 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 11 | 6 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 15 | 15 | 9 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 3 | 1 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 13 | 12 | 12 | 0 | 0 | 0
Vision blurred (Eye disorders) | 3 | 1 | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 6 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.